CLINICAL TRIAL: NCT02229617
Title: A Pilot Study of Subcutaneous vs. Intramuscular Testosterone for Gender Affirming Therapy
Brief Title: Subcutaneous Testosterone Project
Acronym: STP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-00862
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Gender Dysphoria
Keywords: Intramuscular testosterone; Subcutaneous testosterone
MeSH Terms: conditions — Gender Dysphoria | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injectable testosterone (Active Comparator): We will take a group of transgender males, already on a stable dosage of intramuscular testosterone, and then using their same type and dosage, switch them to the subcutaneous injection route. Weekly trough (just before their weekly injection) levels of total serum testosterone will be taken to compare the steady states of those two injection routes.
  Interventions: Drug: Subcutaneous testosterone

INTERVENTIONS:
Drug: Subcutaneous testosterone
  Other Names: Testosterone cypionate; Testosteron enanthate

SUMMARY:
For people who identify as transgender, there is a strong sense that they were born into the wrong body and that their outward looking body does not match how they truly feel about themselves. They feel male, not female and have always felt that way. There is a great deal of discomfort or dysphoria about looking and feeling female, and there is a strong desire to achieve a more masculine appearance. While surgery, clothing and hair for example, can help a person appear more like a male, many transgender males will want to take testosterone to make them feel and look more masculine.

This usually involves injecting testosterone into a muscle every 1-2 weeks for many years. Intramuscular injections can often be uncomfortable or painful, and requires the patient to be taught how to inject themselves. Or somebody else has to do it. There is a growing trend in some transgender men to give their injection just below the skin or subcutaneously (like insulin in a diabetic), because it is less uncomfortable but we don't really know if testosterone gets into the blood in the same way. At least one clinic in the US already suggests that patients can use the subcutaneous method but there is almost no research to show it's the same as intramuscular.

Our project will be looking at a small group of transgender males who are already on intramuscular testosterone and then switch them over to the same dose of subcutaneous testosterone, and then compare their levels of testosterone. If those levels are similar, then patients may chose the less uncomfortable subcutaneous injection.

DETAILED DESCRIPTION:
Rationale:

In caring for transgender males (born female but identify as male), intramuscular (IM) testosterone is considered standard of care if they elect therapy to transition. Yet, IM testosterone has limitations: discomfort; a modest amount of teaching; bleeding concerns if the patient is on anticoagulants; and fluctuations in circulating serum testosterone. Erratic absorption may also led to variability in mood and energy. Due to these limitations, there is a trend, especially in younger patients, to use the more comfortable subcutaneous (SC) route. However, there are little data suggesting equivalency of SC to IM testosterone and virtually no data in transgender males.

Hypothesis:

In transgender males, SC testosterone will yield similar pharmacokinetics and better tolerability when compared to IM testosterone.

Objectives:

1. To validate, using a cross-over design, whether pharmacokinetic parameters of SC vs. IM testosterone administration are similar.
2. To characterize, using a validated pain questionnaire and patient diary, tolerability of SC vs. IM testosterone.

Research Plan:

Patients (19-59 years old) on a weekly self-injection schedule of either T cypionate or enanthate will be included. Patients with medical instability, recent or imminent surgery will be excluded. Twenty-five patients will be recruited from the 6 local Vancouver Coastal HealthTrans Primary Care physicians' clinics.

Using a cross-over design, trough serum testosterone levels from the IM technique will be determined weekly for 3 weeks. Patients will then switch to SC injection of the same testosterone ester and dosage, and weekly trough levels measured for another 8 weeks. These trough measurements will allow us to determine attainment of steady-state testosterone levels. During the 3rd and 11th week, serial testosterone levels will be collected to generate noncompartmental pharmacokinetic parameters, which will be compared between the two techniques. Patients will complete a validated pain analogue questionnaire during the initial 3-week IM phase, and again during weeks 2 and 8 of the SC phase and maintain a diary throughout the study. Descriptive and inferential statistics will be used with p<0.05 denoting significance.

Significance: If SC testosterone yields similar pharmacokinetics and better tolerability than IM testosterone, it will reduce the perceived barrier of IM injections and mitigate non-compliance. There are potential cost savings as patients will not require a clinician to inject. The findings may also be generalized to hypogonadal males. Ultimately, results are crucial to designing a larger multi-center study to provide definitive dosing recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Transgender males or identifying along the male spectrum
* Currently on stable doses of weekly IM testosterone
* Using either Testosterone cypionate or enanthate
* Between 19-59 years old
* Stable doses of regular medications
* Receive their transgender care from one of five(5) Vancouver-based physicians who specialize in transgender care (Three Bridges or Raven Song Community Health Centres).

Exclusion Criteria:

* Medically or psychiatrically unstable
* Recent or imminent surgery (6-8 weeks) that has or may affect testosterone dosage
* Unable to present for nine(9) weeks of weekly blood work and two(2) weeks of alternate day blood work

Ages: 19 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Serum Testosterone (Total) | 11 weeks
  To compare the steady state levels of total serum testosterone using the Subcutaneous (SC) and Intramuscular (IM) injection routes in a group of transgender males who are already on stable IM dosages.

SECONDARY OUTCOMES:
Pharmacokinetics of serum testosterone | 2 weeks
  We will be measuring alternate day serum testosterone levels during the subjects final week of IM testosterone injections (week #3) and the final week of SC testosterone injections (week #11).

OTHER OUTCOMES:
Tolerability and discomfort assessment | 11 weeks
  Study participants will complete a weekly questionnaire regarding tolerability and discomfort, as well as a final questionnaire asking for preferred method of injection.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ensom, Pharm D/PhD, Study Director — University of British Columbia, Faculty of Pharmaceutical Sciences
Locations (2):
- Canada (2):
  - Three Bridges Community Health Centre, Vancouver, British Columbia
  - Raven Song Community Health Centre, Vancouver, British Columbia